CLINICAL TRIAL: NCT01596621
Title: An Open-Label Study to Evaluate Bendamustine Hydrochloride in the Treatment of Chinese Patients With Indolent Non-Hodgkin Lymphoma (NHL) Refractory to Rituximab Treatment
Brief Title: A Study of Bendamustine in the Treatment of Chinese Participants With Indolent Non-Hodgkin Lymphoma Refractory to Rituximab Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/3076
Record Dates: First submitted 2012-05-02; First posted 2012-05-11 (Estimated); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Bendamustine hydrochloride; CEP-18083; Treanda®; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bendamustine (Experimental): Participants will receive bendamustine hydrochloride administered at 120 milligrams (mg)/square meter (m^2) intravenously (IV) as a 60-minute infusion, and not more than 120 minutes, on Days 1 and 2 in each 21-day treatment cycle for 6 planned cycles and up to 8 total cycles.
  Interventions: Drug: Bendamustine hydrochloride

INTERVENTIONS:
Drug: Bendamustine hydrochloride — Bendamustine will be be administered per dose and schedule specified in the arm description.
  Other Names: Treanda®

SUMMARY:
The primary objective of the study is to determine the overall response rate (ORR), which includes complete response (CR) and partial response (PR), to bendamustine treatment in participants with indolent non-Hodgkin lymphoma (NHL) that has progressed after rituximab or a rituximab-containing therapy.

DETAILED DESCRIPTION:
This is a multicenter, nonrandomized, open-label, single-agent clinical study conducted in China, and is designed to investigate the use of bendamustine in the treatment of Chinese participants with relapsed, rituximab-refractory indolent NHL. The study consists of a screening period of up to 4 weeks, a treatment period of approximately 24 weeks (up to eight 21-day cycles), and a long-term follow-up period for up to 2 years after the last dose of study drug. Participants are expected to participate in this study for approximately 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

- The participant has documented relapse from indolent B-cell NHL. Participants with the following subtypes of indolent NHL are eligible for this study: i) small lymphocytic lymphoma (peripheral B cell count <5000 cells/cubic millimeters [mm^3]) ii) lymphoplasmacytic lymphoma iii) splenic marginal zone B-cell lymphoma (±villous lymphocytes) iv) extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue type v) nodal marginal zone lymphoma (±monocytoid B-cells) vi) follicle center lymphoma vii) follicular (grade 1, 2, or 3a) lymphoma

- The participant has disease documented to have progressed despite rituximab treatment. The participant's disease is considered to be rituximab refractory if any of the following criteria are met at any time during the participant's treatment history (progression must be documented by computed tomography [CT] scan or magnetic resonance imaging [MRI] or biopsy) or if a participant has palpable lymph nodes that were well documented in size and, after rituximab treatment, palpable disease remains or comes back [CT, MRI, or biopsy is preferred and performed whenever possible to document progressive disease (PD)]: i) rituximab-only regimen: Participants who receive a full course of single-agent rituximab (at least 2 doses of 375 mg/m^2 [or a therapeutically-active dose] weekly) and have no response (do not obtain a PR or better) to treatment or progress after a full regimen of rituximab was given.

ii) rituximab maintenance therapy or extended schedule: Participants who have a history of a full course of rituximab (at least 2 doses of 375 mg/m^2 [or a therapeutically-active dose] as a single agent [weekly] or in combination with chemotherapy [day 1 of each of 4 cycles]) and are on a maintenance regimen, and progress before the next scheduled rituximab dose or after completing a maintenance rituximab regimen.

iii) rituximab-chemotherapy combination regimen: Participants who receive a full course of rituximab (at least 2 doses of 375 mg/m^2 or a therapeutically-active dose [on day 1 of each of 2 cycles]) in combination with chemotherapy and have no response (do not obtain a PR or better) to treatment or progress after the last dose of rituximab in a regimen.

iv) full rituximab exposure treatment: Participants who have a history of a full course of rituximab treatment (at least 2 doses of 375 mg/m^2 [or a therapeutically-active dose] as a single agent or in combination with chemotherapy) and, in a subsequent rituximab/chemotherapy combination regimen, have no response (do not obtain a PR or better) to treatment or progress after the last dose of rituximab in a given regimen, even if the subsequent regimen included less than 2 doses of rituximab. Participants could receive additional systemic treatment after the qualifying rituximab regimen.

* The participant has received treatment with at least 1, but no more than 3, previous chemotherapy regimens. A regimen is defined as a new treatment combination or agent. Retreatment with the identical regimen or agent does not count as a new regimen; however, change from cyclophosphamide, vincristine, and prednisolone (CVP) to cyclophosphamide, doxorubicin, vincristine, and prednisolone (CHOP) is counted as a new regimen. Rituximab, radioimmunotherapy, or other biologic treatments not combined with chemotherapy are not counted as a regimen.
* The participant has a bidimensionally measurable disease with at least 1 lesion measuring 2.0 centimeters (cm) or more in a single dimension. Participants who have previous involved-field irradiation can be included, provided the irradiated area is not the only source of measurable disease.
* The participant has a World Health Organization (WHO) performance status of 0, 1, or 2.
* The participant has absolute neutrophil count (ANC) 1000 cells/mm^3 or more and platelet count 85000 cells/mm^3 or more.
* The participant has a creatinine clearance of more than 30 mL/min as determined by the Cockcroft-Gault calculation.
* The participant has adequate hepatic function (no more than 2.5 times the upper limit of normal (ULN) for aspartate aminotransferase (AST) and alanine aminotransferase (ALT), and no more than 1.5 times the upper limit of the normal range (ULN) for total bilirubin). Participants with nonclinically significant elevations of bilirubin due to Gilbert's disease are eligible.
* The participant has had a bone marrow biopsy within 6 weeks before the 1st dose of bendamustine.
* Women of childbearing potential (not surgically sterile or 1 year postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method starting 2 weeks before the start of study drug treatment, during study drug treatment, and for 3 months after the end of study drug treatment. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* Women of childbearing potential must have a negative serum or urine pregnancy test.
* Men not surgically sterile or who are capable of producing offspring must practice abstinence or use a barrier method of birth control, and must agree to continue use of this method starting 2 weeks before the start of study drug treatment, during study drug treatment, and for 3 months after the end of study drug treatment.
* The participant has an estimated life expectancy of at least 3 months.
* The participant (or participant's legal representative) provides written informed consent.

Exclusion Criteria:

* The participant has received previous radiotherapy, radioimmunotherapy, chemotherapy, or immunotherapy within 4 weeks before day 1 of cycle 1 or has failed to recover (to Common Terminology Criteria for Adverse Events [CTCAE] toxicity grade 1 or 2) from clinically significant nonhematologic adverse events due to any agents administered previously.
* The participant has received treatment with an investigational agent within 4 weeks of day 1 of cycle 1.
* The participant has received hematopoietic growth factors within 4 weeks of day 1 of cycle 1. However, participants receiving chronic erythropoietin treatment are eligible for inclusion in this study.
* The participant has a history of previous high-dose chemotherapy with allogeneic stem cell support (history of autologous stem cell support is permissible).
* The participant is receiving or has received treatment with therapeutic doses of systemic steroids within 4 weeks of day 1 of cycle 1. (Low doses of chronic steroids [prednisone or equivalent] up to 20 mg/day for non-neoplastic disorders or for indications other than lymphoma or lymphoma-related complications are permitted.)
* The participant has transformed disease.
* The participant has any history of central nervous system (CNS) or leptomeningeal lymphoma.
* The participant has, or has had within the past 5 years, an active malignancy other than the target cancer. The exceptions are prostate cancer (Gleason grade <6 with prostate specific antigen [PSA] levels within the normal range), in situ cervical or breast carcinoma, and nonmelanoma skin cancer that have received definitive treatment.
* The participant is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study immediately.)
* The participant has a serious infection, medical condition, or psychiatric condition that, in the opinion of the investigator, might interfere with the achievement of the study objectives.
* The participant is known to be positive for human immunodeficiency virus (HIV), have active hepatitis B, or active hepatitis C (anti-hepatitis C virus [HCV] positive). Hepatitis B surface antigen must be tested. The determination of active disease is left up to the Investigator.
* The participant has a known hypersensitivity to mannitol.
* The participant has used bendamustine previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2015-06-18 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (27):
- China (27):
  - Teva Investigational Site 001, Beijing
  - Teva Investigational Site 026, Beijing
  - Teva Investigational Site 022, Beijing
  - Teva Investigational Site 004, Beijing
  - Teva Investigational Site 003, Beijing
  - Teva Investigational Site 002, Beijing
  - Teva Investigational Site 023, Beijing
  - Teva Investigational Site 016, Beijing
  - Teva Investigational Site 021, Beijing
  - Teva Investigational Site 015, Changchun
  - Teva Investigational Site 010, Chengdu
  - Teva Investigational Site 008, Guangzhou
  - Teva Investigational Site 007, Guangzhou
  - Teva Investigational Site 011, Hangzhou
  - Teva Investigational Site 019, Harbin
  - Teva Investigational Site 025, Hefei
  - Teva Investigational Site 024, Lanzhou
  - Teva Investigational Site 012, Nanjing
  - Teva Investigational Site 013, Nanjing
  - Teva Investigational Site 006, Shanghai
  - Teva Investigational Site 005, Shanghai
  - Teva Investigational Site 009, Shenyang
  - Teva Investigational Site 027, Shenyang
  - Teva Investigational Site 020, Suzhou
  - Teva Investigational Site 014, Tianjin
  - Teva Investigational Site 018, Xi'an
  - Teva Investigational Site 017, Zhengzhou

REFERENCES:
- [Derived] Shi YK, Hong XN, Yang JL, Xu W, Huang HQ, Xiao XB, Zhu J, Zhou DB, Han XH, Wu JQ, Zhang MZ, Jin J, Ke XY, Li W, Wu DP, Yang SM, Du X, Jia YQ, Liu AC, Liu DH, Shen ZX, Zhang LS, James L, Hellriegel E. Bendamustine treatment of Chinese patients with relapsed indolent non-Hodgkin lymphoma: a multicenter, open-label, single-arm, phase 3 study. Chin Med J (Engl). 2021 May 6;134(11):1299-1309. doi: 10.1097/CM9.0000000000001463. PMID 33967195

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine: Participants received bendamustine hydrochloride administered at 120 milligrams (mg)/square meter (m^2) intravenously (IV) as a 60-minute infusion, and not more than 120 minutes, on Days 1 and 2 in each 21-day treatment cycle for 6 planned cycles and up to 8 total cycles.
Period: Overall Study
Arm/Group | Bendamustine
Started | 102
Received at Least 1 Dose of Study Drug | 102
Completed | 24
Not Completed | 78
Not completed — Death | 4
Not completed — Withdrawal by Subject | 9
Not completed — Disease Progression | 49
Not completed — Lost to Follow-up | 3
Not completed — Other than specified | 13

BASELINE CHARACTERISTICS:
Population: The primary analysis set (PAS) included all enrolled participants who were treated with any amount of study drug.
Groups:
- Bendamustine: Participants received bendamustine hydrochloride administered at 120 mg/m^2 IV as a 60-minute infusion, and not more than 120 minutes, on Days 1 and 2 in each 21-day treatment cycle for 6 planned cycles and up to 8 total cycles.
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 102

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) (Assessed by Independent Review Committee [IRC])
Description: The ORR was defined as the percentage of participants who achieved a best response of complete response (CR) or partial response (PR) during the study based on the modified International Workshop Response Criteria. CR: disappearance of all evidence of disease; nodal masses regression on normal size on computed tomography (CT); spleen and liver not palpable and nodule disappeared; bone marrow infiltrate cleared on repeat biopsy. PR: Regression of measurable disease and no new sites; nodal masses ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 largest dominant masses and no increase in size of other nodes; spleen and liver ≥50% decrease in SPD of nodules and no increase in size of liver or spleen.
Time Frame: From the date of the first administration of bendamustine to the first documentation of disease progression/relapse, new anticancer therapy, or death (regardless of cause), whichever occurred first (up to 2.5 Years)
Population: The primary analysis set (PAS) included all enrolled participants who were treated with any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
percentage of participants | 73

2. Secondary Outcome: Duration of Response (DOR) (Assessed by IRC)
Description: Duration of response was defined as the time from the date of first documentation of response to the first documentation of disease progression, new anticancer therapy, or death (regardless of cause), whichever occurred first for participants with a best response of CR or PR determined by the modified International Workshop Response Criteria. CR: disappearance of all evidence of disease; nodal masses regression on normal size on CT; spleen and liver not palpable and nodule disappeared; bone marrow infiltrate cleared on repeat biopsy. PR: Regression of measurable disease and no new sites; nodal masses ≥50% decrease in SPD of up to 6 largest dominant masses and no increase in size of other nodes; spleen and liver ≥50% decrease in SPD of nodules and no increase in size of liver or spleen. Disease progression: any new lesion or increase by ≥50% of previously involved sites from nadir.
Time Frame: From the date of first documentation of response to the first documentation of disease progression, new anticancer therapy, or death (regardless of cause), whichever occurred first (up to 2.5 Years)
Population: The PAS included all enrolled participants who were treated with any amount of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine
Number analyzed (Participants) | 74
months | 16.2 [9.3 to NA] — Due to smaller number of participants with an event the upper limit of 95% confidence interval (CI) could not be calculated.

3. Secondary Outcome: Progression-Free Survival (Assessed by IRC)
Description: Progression free survival was defined as the time from the date of the first administration of bendamustine to the first documentation of disease progression/relapse, new anticancer therapy, or death (regardless of cause), whichever occurred first for all participants. Disease progression/relapse: appearance of any new lesion or increase by ≥50% of previously involved sites from nadir.
Time Frame: as for outcome 1
Population: The PAS included all enrolled participants who were treated with any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
months | 18.6 [12.3 to NA] — Due to smaller number of participants with an event the upper limit of 95% CI could not be calculated.

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bendamustine
Time Frame: Prior to the start of infusion on Day 1 for up to 24 hours after the end of infusion during Cycle 1 (each cycle is 21 days)
Population: The pharmacokinetic analysis set included all enrolled participants who were treated with any amount of study drug and for whom at least 1 pharmacokinetic parameter was calculated.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliters (mL)
Arm/Group | Bendamustine
Number analyzed (Participants) | 15
nanograms (ng)/milliliters (mL) | 3909.9 (2995.83)

5. Secondary Outcome: Time to Reach Cmax (Tmax) of Bendamustine
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Bendamustine
Number analyzed (Participants) | 15
hours | 1.30 [0.58 to 1.97]

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Drug Concentration (AUC0-t) of Bendamustine
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Bendamustine
Number analyzed (Participants) | 15
ng*hour/mL | 5660.7 (3932.45)

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUC0-∞) of Bendamustine
Time Frame: as for outcome 4
Population: The pharmacokinetic analysis set included all enrolled participants who were treated with any amount of study drug and for whom at least 1 pharmacokinetic parameter was calculated. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Bendamustine
Number analyzed (Participants) | 10
ng*hour/mL | 6278.7 (4724.82)

8. Secondary Outcome: Rate Constant for Elimination (λz) of Bendamustine
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Bendamustine
Number analyzed (Participants) | 10
1/hour | 0.4525 (0.24245)

9. Secondary Outcome: Percentage of the AUC0-∞ Based on Extrapolation (%AUCext)
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of AUC0-∞
Arm/Group | Bendamustine
Number analyzed (Participants) | 10
percentage of AUC0-∞ | 0.01 (0.004)

10. Secondary Outcome: Half-Life (t½) of Bendamustine
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bendamustine
Number analyzed (Participants) | 10
hours | 1.83 (0.684)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first administration of bendamustine through 30 days after the last administration (up to 2.5 Years)
Population: Safety analysis set included all enrolled participants who were treated with any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
Participants | 101

12. Secondary Outcome: World Health Organization (WHO) Performance Status
Description: Number of participants with WHO performance status (improved, stayed the same, and deteriorated) at the end of treatment have been reported.
Time Frame: At the end of treatment (up to 2.5 years)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 86
Participants
  Improved | 6
  Stayed the same | 73
  Deteriorated | 7

13. Secondary Outcome: Number of Participants Who Need At Least 1 Hematologic Supportive Care (Plasma, Blood Cells, or Cytokines)
Time Frame: From first administration of bendamustine up to the end of treatment (up to 2.5 Years)
Population: The PAS included all enrolled participants who were treated with any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
Participants | 71

14. Secondary Outcome: Number of Participants With Concomitant Medication Usage
Description: Concomitant medications included all medications taken while the participant received study drug.
Time Frame: From first administration of bendamustine up to the end of treatment (up to 2.5 Years)
Population: Safety analysis set included all enrolled participants who were treated with any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 102
Participants | 102

ADVERSE EVENTS:
Time Frame: From first administration of bendamustine through 30 days after the last administration (up to 2.5 Years)
Description: Safety analysis set included all enrolled participants who were treated with any amount of study drug.
Arm/Group | Bendamustine
Serious Adverse Events (participants affected / at risk) | 30/102
Other Adverse Events (participants affected / at risk) | 99/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=102)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Hepatitis B (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 1 (2)
White blood cell count increased (Investigations) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=102)
Anaemia (Blood and lymphatic system disorders) | 26 (91)
Leukopenia (Blood and lymphatic system disorders) | 46 (235)
Lymphopenia (Blood and lymphatic system disorders) | 11 (44)
Neutropenia (Blood and lymphatic system disorders) | 47 (263)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (79)
Nausea (Gastrointestinal disorders) | 45 (110)
Vomiting (Gastrointestinal disorders) | 32 (81)
Asthenia (General disorders) | 15 (20)
Fatigue (General disorders) | 8 (13)
Infusion site phlebitis (General disorders) | 13 (18)
Pyrexia (General disorders) | 24 (43)
Upper respiratory tract infection (Infections and infestations) | 11 (17)
Alanine aminotransferase increased (Investigations) | 14 (21)
Aspartate aminotransferase increased (Investigations) | 10 (15)
Haemoglobin decreased (Investigations) | 11 (35)
Lymphocyte count decreased (Investigations) | 20 (69)
Neutrophil count decreased (Investigations) | 47 (247)
Platelet count decreased (Investigations) | 41 (136)
Weight decreased (Investigations) | 10 (12)
White blood cell count decreased (Investigations) | 55 (283)
Decreased appetite (Metabolism and nutrition disorders) | 26 (62)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (15)
Rash (Skin and subcutaneous tissue disorders) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.